CLINICAL TRIAL: NCT01035229
Title: A Randomized Phase III, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Everolimus (RAD001) in Adult Patients With Advanced Hepatocellular Carcinoma After Failure of Sorafenib Treatment - The EVOLVE-1 Study
Brief Title: Global Study Looking at the Combination of RAD001 Plus Best Supportive Care (BSC) and Placebo Plus BSC to Treat Patients With Advanced Hepatocellular Carcinoma.
Acronym: EVOLVE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAD001O2301; 2009-010196-25 (EudraCT Number)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Carcinoma
Keywords: Hepatocellular carcinoma; randomized trial; medical treatment; RAD001; placebo; Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus + Best Supportice Care (BSC) (Experimental): Patients were assigned to the Everolimus + BSC arm in a ratio of 2:1 over the Placebo arm. Everolimus was taken as a daily oral dose of 7.5 mg and was defined as the investigational drug. In addition to taking Everolimus, all patients also received BSC as per normal local practice.
  Interventions: Drug: Everolimus; Other: Best Supportive Care (BSC)
- Placebo + Best Supportive Care (Placebo Comparator): Placebo Everolimus was taken as a daily oral dose of 7.5 mg and was defined as the control drug. In addition to taking Placeb Everolimus, all patients also received BSC as per normal local practice.
  Interventions: Drug: Everolimus Placebo; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Everolimus — Everolimus (labeled as RAD001) was formulated as tablets of 2.5 mg strength and blisterpacked in units of 10 tablets.
  Other Names: RAD001
  Arms: Everolimus + Best Supportice Care (BSC)
Drug: Everolimus Placebo — Everolimus Placebo matched to the everolimus 2.5 mg tablet strength was blister-packed in units of 10 tablets. Matching placebo tablets were formulated to be indistinguishable from the everolimus tablets. Everolimus placebo was taken as a daily oral dose of 7.5 mg and was defined as the control drug.
  Arms: Placebo + Best Supportive Care
Other: Best Supportive Care (BSC) — BSC was defined as drug or non-drug therapies, nutritional support, physical therapy or anything that the Investigator believed to be in the patient's best interest, but excluding other antineoplastic treatments. BSC administered to the patient throughout the study was to be reported on the Concomitant Medication/Significant Non-Drug Therapy electronic case report from (eCRF). Permitted BSC treatments during the study included, but were not limited to, the following: Pain medication to allow the patient to be as comfortable as possible, Bisphosphonates for bone metastases, Localized radiotherapy, for the treatment of pre-existing, painful bone metastases, Nutritional support or appetite stimulants (i.e. megestrol) as recommended by the Investigator, Oxygen therapy and blood products or transfusions

SUMMARY:
The purpose of this study is to compare treatment with RAD001 plus best supportive care (BSC) to placebo plus BSC in patients with advanced HCC whose disease progressed while on or after sorafenib treatment or who are intolerant to sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Advanced liver cancer
* Prior systemic treatment with sorafenib for advanced HCC and for whom their disease progressed during or after sorafenib treatment, or were intolerant to sorafenib treatment. Specifically, this can be defined as:

  * Documented radiological confirmation (radiology scans or report) of disease progression during or after sorafenib treatment
  * Intolerance to sorafenib (at any dose and/or duration) is defined as documented sorafenib-related grade 3 or 4 adverse events that led to sorafenib discontinuation.

NOTE:

* Sorafenib must be the last antineoplastic treatment before randomization
* Prior local and/or hormonal therapy (e.g., tamoxifen) before sorafenib is allowed
* One systemic chemotherapy regimen for advanced HCC is allowed before sorafenib treatment

  * ECOG performance status of ≤ 2
  * Child-Pugh A

Exclusion Criteria:

* Active bleeding during the last 28 days
* Prior therapy with mTOR inhibitors
* Prior liver or other organ transplantation which mandates systemic immunosuppression

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (122):
- United States (19):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Compassionate Cancer Care Medical Group CCCMG, Fountain Valley, California
  - University of California San Diego - Moores Cancer Center SC - 3, La Jolla, California
  - California Pacific Medical Center California Pacific Med, San Francisco, California
  - Rocky Mountain Cancer Centers RMCC - Denver-Midtown (4), Greenwood Village, Colorado
  - Queen's Medical Center Queens Cancer Center, Honolulu, Hawaii
  - The Sidney Kimmel Cancer Center at Johns Hopkins Hospital Dept. of SKCC @ JHU, Baltimore, Maryland
  - Massachusetts General Hospital Dept. of Mass General Hospital, Boston, Massachusetts
  - Midwest Cancer Care Physicians Research Medical Center, Kansas City, Missouri
  - VA Sierra Nevada Health Care System Dept. of VA Sierra Nevada HCS, Reno, Nevada
  - University of Rochester Medical Center Rochester, Rochester, New York
  - Northwest Cancer Specialists Rose Quarter Cancer Center, Portland, Oregon
  - St. Luke's Hospital and Health Network St. Luke's Cancer Network (2), Bethlehem, Pennsylvania
  - Texas Cancer Center - Abilene, Abilene, Texas
  - Methodist Charlton Cancer Center Methodist, Dallas, Texas
  - University of Texas Southwestern Medical Center DeptofSimmons Cancer Center(3), Dallas, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio, San Antonio, Texas
  - Blue Ridge Research Center at Roanoke Neurological Center Blue Ridge Cancer Care, Roanoke, Virginia
  - University of Washington Cancer Care SC, Seattle, Washington
- Australia (5):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (6):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- France (18):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen Cedex9
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille Cédex 5
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
- Germany (11):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Greece (3):
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- Israel (2):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (13):
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Frattamaggiore
  - Novartis Investigative Site, Napoli
- Japan (17):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (5):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
- Taiwan (7):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Liouying Township
- Novartis Investigative Site, Bangkok, Thailand

REFERENCES:
- [Derived] Zhu AX, Chen D, He W, Kanai M, Voi M, Chen LT, Daniele B, Furuse J, Kang YK, Poon RT, Vogel A, Chiang DY. Integrative biomarker analyses indicate etiological variations in hepatocellular carcinoma. J Hepatol. 2016 Aug;65(2):296-304. doi: 10.1016/j.jhep.2016.04.015. Epub 2016 Apr 27. PMID 27130844
- [Derived] Zhu AX, Kudo M, Assenat E, Cattan S, Kang YK, Lim HY, Poon RT, Blanc JF, Vogel A, Chen CL, Dorval E, Peck-Radosavljevic M, Santoro A, Daniele B, Furuse J, Jappe A, Perraud K, Anak O, Sellami DB, Chen LT. Effect of everolimus on survival in advanced hepatocellular carcinoma after failure of sorafenib: the EVOLVE-1 randomized clinical trial. JAMA. 2014 Jul 2;312(1):57-67. doi: 10.1001/jama.2014.7189. PMID 25058218
- See also: Related Info — https://www.novartisclinicaltrials.com/TrialConnectWeb/home.nov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 763 patients screened, 546 randomized. At 14Jun2013 data cut-off (final analysis), 3 pts in everolimus arm, 6 in placebo arm were still on treatment. Of 9 pts, 3 receiving placebo discontinued due to disease progression. Remaining 6 completed study due to sponsor's decision to end study after final results. The LPLV was 15Oct2013.
Groups:
- Everolimus + Best Supportive Care (BSC): Patients were assigned to the Everolimus + BSC arm in a ratio of 2:1 over the Placebo arm. Everolimus was taken as a daily oral dose of 7.5 mg but dose adjustments of study drug (reduction, interruption or possible dose re-escalation to starting dose) according to safety findings were allowed. In addition to taking Everolimus, all patients also received BSC as per normal local practice.
- Placebo + Best Supportive Care: Placebo-Everolimus was taken as a daily oral dose of 7.5 mg and was defined as the control drug. In addition to taking Placebo Everolimus, all patients also received BSC as per normal local practice.
Period: Overall Study
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Started | 362 | 184
Completed | 0 | 0
Not Completed | 362 | 184
Not completed — Adverse Event | 61 | 14
Not completed — Withdrawal by Subject | 20 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 1 | 1
Not completed — Death | 13 | 5
Not completed — New cancer therapy | 2 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Sponsor's decision to end study | 3 | 3
Not completed — Disease Progression | 261 | 152

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care | Total
Number analyzed (Participants) | 362 | 184 | 546
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (11.70) | 64.2 (10.41) | 64.8 (11.28)
Age, Customized [Number; unit: Participants]
  < 35 years | 7 | 1 | 8
  >=35 - <55 years | 48 | 31 | 79
  >=55 - <65 years | 100 | 61 | 161
  >= 65 years | 207 | 91 | 298
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 24 | 83
  Male | 303 | 160 | 463
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 192 | 110 | 302
  Black | 6 | 3 | 9
  Asian | 137 | 58 | 195
  Pacific Islander | 0 | 1 | 1
  Other | 27 | 12 | 39
Weight [Mean (Standard Deviation); unit: kg] | 69.6 (15.62) | 71.3 (17.71) | 70.2 (16.35)
Height [Mean (Standard Deviation); unit: cm] | 167.9 (8.66) | 169.2 (8.84) | 168.3 (8.73)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.5 (4.64) | 24.8 (4.99) | 24.6 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. The comparison of OS between the 2 arms was done using a stratified log-rank test at one-sided 2.5% level of significance.
Time Frame: When 454 OS events were observed
Population: The Full Analysis Set (FAS) comprised all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Number analyzed (Participants) | 362 | 184
Months | 7.56 [6.70 to 8.74] | 7.33 [6.28 to 8.74]

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the date of the first documented radiologic confirmation of disease progression. Since the study did not meet the primary objective, TTP was not formally tested.
Time Frame: Until all patients have disease progression or leave study due to intolerable adverse events- Estimate of 1 year for each patient
Population: The Full Analysis Set (FAS) comprised all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Number analyzed (Participants) | 362 | 184
Months | 2.96 [2.79 to 4.01] | 2.60 [1.48 to 2.83]

3. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: DCR is defined as the proportion of participants with a best objective response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) according to RECIST. The BOR was the best response recorded from the start of the treatment until disease progression. CR is disappearance of all target lesions; PR is at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters; SD is neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD. PD is at least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: as for outcome 2
Population: The Full Analysis Set (FAS) comprised all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Number analyzed (Participants) | 362 | 184
Percentage of Participants | 56.1 | 45.1

4. Secondary Outcome: Time to Definitive Deterioration of ECOG Performance Score (PS) Score
Description: Change in Eastern Cooperative Oncology Group (ECOG) were assessed by time to definitive performance status deterioration by at least one category on the ECOG scale. Deterioration was considered definitive if no improvement in the ECOG PS was observed at a subsequent measurement. ECOG PS: 0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair; 5=Dead
Time Frame: as for outcome 2
Population: The Full Analysis Set (FAS) comprised all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Number analyzed (Participants) | 362 | 184
Months | 4.27 [3.32 to 4.86] | 4.47 [3.02 to 6.08]

5. Secondary Outcome: Time to Definitive Deterioration of EORTC QLQ-C30 Scores
Description: The primary quality of life endpoint was the time to definitive 5% deterioration from baseline in the global health status/quality of life scale of the EORTC QLQ-C30 questionnaire. Definitive deterioration by at least 5% is defined as a decrease in score by at least 5% compared to baseline, with no later observed increase above this threshold. The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the healthrelated quality of life (QoL) of cancer patients participating in international clinical trials. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time Frame: Until all patients have disease progression or leave study due to intolerable adverse events - Estimate of 1 year for each patient.
Population: The Full Analysis Set (FAS) comprised all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Number analyzed (Participants) | 362 | 184
Months | 2.86 [2.66 to 4.11] | 3.45 [2.79 to 4.17]

6. Secondary Outcome: Pharmacokinetics Assessments - Cmin
Description: Cmin is the pre-dose blood concentration at steady-state (ng/mL). Pre-dose (Cmin) blood samples were collected from all patients in both arms at Visit 3. Steady-state for the Cmin sample was defined as continuous administration of the same dose in the last 4 days prior to the collection of the Cmin sample. Steady-state for the 5 mg every other day regimen was defined as the state when the 5 mg dose was taken 2 days and 4 days before sampling. PK samples were only drawn at visit 3, and only analyzed for patients receiving everolimus at steady state (if patients had received the dose the previous 4 days). In addition summary statistics were only done for each everolimus dose when 3 samples were available. Only valid pre-dose (Cmin) everolimus samples were included in the analysis.
Time Frame: as for outcome 5
Population: Safety Set consisted of all patients who received at least one dose of study treatment with a valid postbaseline assessment. All PK analyses were based on the Safety Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus 7.5mg + Best Supportive Care (BSC): Patients were assigned to the Everolimus + BSC arm in a ratio of 2:1 over the Placebo arm. Everolimus was taken as a daily oral dose of 7.5 mg but dose adjustments of study drug (reduction, interruption or possible dose re-escalation to starting dose) according to safety findings were allowed. In addition to taking Everolimus, all patients also received BSC as per normal local practice.
- Everolimus 5mg + Best Supportive Care (BSC): Everolimus was taken as a daily oral dose of 7.5 mg but dose adjustments of study drug (reduction, interruption or possible dose re-escalation to starting dose) according to safety findings were allowed.
Arm/Group | Everolimus 7.5mg + Best Supportive Care (BSC) | Everolimus 5mg + Best Supportive Care (BSC)
Number analyzed (Participants) | 206 | 10
ng/mL | 16.141 (9.2297) | 9.318 (4.9705)

7. Secondary Outcome: Pharmacokinetics Assessments - Cmax
Description: Cmax is the maximum (peak) blood drug concentration after dose administration (ng/mL) calculated as the maximum of C1h and C2h. C1h was 1 hour post-dose blood concentration (ng/mL) and C2h was 2 hour post-dose blood concentration (ng/mL). C1h and C2h post-dose samples were collected from all patients in both arms at Visit 3. Steady-state for the C1h and C2h samples was defined as continuous administration of the same dose in the previous 4 days and the day on which the C1h and C2h samples were collected. Steady-state for the 5 mg every other day regimen was defined as the state when the 5 mg dose was taken 2 days and 4 days before sampling. PK samples were only drawn at visit 3, and only analyzed for patients receiving everolimus at steady state (if patients had received the dose the previous 4 days). In addition summary statistics were only done for each everolimus dose when 3 samples were available. Only valid C1h and C2h everolimus samples were included in the analysis.
Time Frame: as for outcome 2
Population: Safety Set consists of all patients who received at least one dose of study treatment with a valid postbaseline assessment. All PK analyses were based on the Safety Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Everolimus 7.5mg + Best Supportive Care (BSC) | Everolimus 5mg + Best Supportive Care (BSC)
Number analyzed (Participants) | 229 | 13
ng/mL | 47.881 (21.0999) | 31.592 (21.1622)

ADVERSE EVENTS:
Description: Three patients (1 in the everolimus arm and 2 in the placebo arm) were excluded from the Safety Set as these patients were randomized but never received any study treatment.
Arm/Group | Everolimus + Best Supportive Care (BSC) | Placebo + Best Supportive Care
Serious Adverse Events (participants affected / at risk) | 171/361 | 64/182
Other Adverse Events (participants affected / at risk) | 343/361 | 147/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Best Supportive Care (BSC) (N=361) | Placebo + Best Supportive Care (N=182)
Anaemia (Blood and lymphatic system disorders) | 14 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 8
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 13 | 11
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2
Ileal ulcer (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 3
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 9 | 3
Chills (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 5 | 4
Hyperpyrexia (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 4 | 2
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 14 | 2
Sudden death (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 8 | 3
Hepatic failure (Hepatobiliary disorders) | 5 | 4
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 5
Jaundice (Hepatobiliary disorders) | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Allergic oedema (Immune system disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial toxaemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholangitis suppurative (Infections and infestations) | 1 | 0
Citrobacter infection (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Listeriosis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Morganella infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 4 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 18 | 1
Sepsis (Infections and infestations) | 6 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0
C-reactive protein abnormal (Investigations) | 1 | 0
Cardiac enzymes increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 2 | 0
Hepatic encephalopathy (Nervous system disorders) | 5 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 3
Disorientation (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 11 | 2
Renal failure acute (Renal and urinary disorders) | 8 | 2
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Immobilisation prolonged (Social circumstances) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 2
Vascular compression (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Best Supportive Care (BSC) (N=361) | Placebo + Best Supportive Care (N=182)
Anaemia (Blood and lymphatic system disorders) | 56 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 2
Abdominal pain (Gastrointestinal disorders) | 54 | 27
Abdominal pain upper (Gastrointestinal disorders) | 28 | 17
Ascites (Gastrointestinal disorders) | 51 | 23
Constipation (Gastrointestinal disorders) | 31 | 23
Diarrhoea (Gastrointestinal disorders) | 94 | 25
Dry mouth (Gastrointestinal disorders) | 23 | 5
Nausea (Gastrointestinal disorders) | 60 | 25
Stomatitis (Gastrointestinal disorders) | 142 | 9
Vomiting (Gastrointestinal disorders) | 55 | 17
Asthenia (General disorders) | 59 | 31
Fatigue (General disorders) | 90 | 30
Oedema peripheral (General disorders) | 100 | 25
Pyrexia (General disorders) | 86 | 13
Hepatitis B (Infections and infestations) | 25 | 8
Alanine aminotransferase increased (Investigations) | 11 | 11
Aspartate aminotransferase increased (Investigations) | 23 | 19
Gamma-glutamyltransferase increased (Investigations) | 18 | 12
Platelet count decreased (Investigations) | 21 | 0
Weight decreased (Investigations) | 34 | 8
Decreased appetite (Metabolism and nutrition disorders) | 114 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 9
Dysgeusia (Nervous system disorders) | 31 | 4
Headache (Nervous system disorders) | 26 | 9
Insomnia (Psychiatric disorders) | 37 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 78 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 19 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 29
Rash (Skin and subcutaneous tissue disorders) | 76 | 16

LIMITATIONS AND CAVEATS:
Three patients (1 in the everolimus arm and 2 in the placebo arm were excluded from the Safety Set. These three patients were randomized but never received any study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.